CLINICAL TRIAL: NCT05448430
Title: iTBS Can Increase Frontal Dopamine Release and Improve Glucose Metabolism in PET Dopamine Imaging of Patients With Schizophrenia.
Brief Title: iTBS Can Increase Frontal Dopamine Release in PET Dopamine Imaging.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: WU2022PETTMS
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- predominant negative symptoms (Experimental): iTBS for predominant negative symptoms
  Interventions: Device: Theta burst stimulation
- positive symptoms (No Intervention)
- healthy control (No Intervention)

INTERVENTIONS:
Device: Theta burst stimulation — a new paradigm of high frequency repetitive transcranial magnetic stimulation
  Arms: predominant negative symptoms

SUMMARY:
Aim: 1. To confirm that patients with predominant negative symptoms in schizophrenia have deficits in frontal cortical dopamine release when compared with healthy control and patients with positive symptoms.

2. Our previous study found patients with negative symptoms have more possibilities to have disorders in glucose metabolism, we wonder whether dopamine release, negative symptoms or glucose metabolism can be improved by iTBS.

Study design: Case control study.

DETAILED DESCRIPTION:
Eligibility Criteria: Predominant negative symptoms for Positive and Negative Syndrome Scale factor score for negative symptoms of 24 or more, and score of 4 or more on at least two of three core negative PANSS items, PANSS for positive symptoms of 19 or less, HAMD depression scale of 16 or less. Predominant positive symptoms for PANSS for positive symptoms of 20 or more. Healthy control will be recruited matching the age and sex of patient groups, Outcome Measures: Oral glucose tolerance test (OGTT), PET dopamine imaging.

ELIGIBILITY:
Inclusion Criteria for negative group

* diagnosed with schizophrenia according to ICD-10 or DSM-V
* Positive and Negative Syndrome Scale factor score for negative symptoms of 24 or moreand score of 4 or more on at least two of three core negative PANSS items
* PANSS for positive symptoms of 19 or less, and HAMD depression scale of 16 or less.
* drug-naive Inclusion Criteria for positive group
* PANSS for positive symptoms of 20 or more
* drug-naive

Exclusion Criteria:

* drug or alcohol addiction
* diagnosed with other major mental disorders according to ICD-10 or DSM-V

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
PET dopamine imaging and OGTT | immediate
  PET dopamine imaging and OGTT after iTBS

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided